CLINICAL TRIAL: NCT02082340
Title: Innovative Approach in Tuberculosis Care in Armenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varduhi Petrosyan (Other)
Collaborators: Grand Challenges Canada (Other); National Tuberculosis Control Center, Ministry of Health, Republic of Armenia (Unknown)
Responsible Party: Sponsor-Investigator, Varduhi Petrosyan, MS, PHD, American University of Armenia Fund
Organization: American University of Armenia Fund (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S5 0399-01_GCC
Record Dates: First submitted 2014-03-04; First posted 2014-03-10 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Armenia; Clinical trial; Directly Observed Therapy (DOT); Self-administered drug intake
MeSH Terms: conditions — Tuberculosis; Directly Observed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): The intervention includes the following components: self-administered drug intake strategy, TB knowledge and socio-psychological counseling session, SMS text messages, phone calls, educational leaflet
  Interventions: Behavioral: TB knowledge and socio-psychological counseling session; Other: SMS text messages; Other: phone calls; Behavioral: Self-administered drug intake strategy; Behavioral: Educational leaflet
- Control arm (No Intervention): patients included in the control arm will receive traditional - clinical Directly Observed Therapy (DOT) as recommended by WHO

INTERVENTIONS:
Behavioral: TB knowledge and socio-psychological counseling session — TB patients and their family members will participate in one-day counseling session provided by a trained psychologist and a TB nurse
  Arms: Intervention arm
Other: SMS text messages — TB patients will receive SMS text messages every morning (except Sunday) during the whole ambulatory TB treatment phase as a reminder for taking the TB medication prescribed and provided by the TB physician
  Arms: Intervention arm
Other: phone calls — Family members of the TB patients will receive phone calls every evening (except Sunday) during the whole ambulatory TB treatment phase to assure that the patient takes the medication prescribed and provided by the TB physician and to collect information on treatment adherence and possible side effects.
  Arms: Intervention arm
Behavioral: Self-administered drug intake strategy — Once a week TB patients will receive the TB medication from their local outpatient TB centers and will use the medication every day (six days a week, except Sunday according to the TB treatment protocol) at home under supervision of a family member in charge.
  Arms: Intervention arm
Behavioral: Educational leaflet — Educational leaflet containing information on TB infection; infection control measures; importance of TB treatment adherence and family support will be provided to all TB patients at the end of the counselling session
  Arms: Intervention arm

SUMMARY:
Randomized trial tests effectiveness of self-administered drug intake by empowered TB patients - supervised by a trained family member and supported by medical counseling and reminders - to improve treatment adherence and treatment success rates, and thereby forestall TB and MDR-TB epidemics.

DETAILED DESCRIPTION:
The innovative treatment approach integrates several educational, technological, and social evidence-based components. The aim of this study is to pilot the innovative approach for drug-sensitive TB patients during the outpatient phase of tuberculosis treatment. To test the effectiveness of the innovative approach (intervention) a randomized controlled trial with two arms will be conducted. The intervention arm will include drug-sensitive tuberculosis patients that are treated according to the innovative approach, which includes self-administered drug intake supervised by a family member, TB patient and family member training (including distribution of a leaflet about TB) and psychological counseling, reminder text messages to TB patients, and reminder phone call to TB patient family members. The control arm will include drug-sensitive tuberculosis patients that receive the regular Directly Observed Therapy recommended by the World Health Organization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of drug-sensitive TB
* Age 18 years old and above
* Understanding and reading in Armenian
* Completion of the intensive treatment phase

Exclusion Criteria:

* Involvement in the Home Based TB Treatment Program of the National TB Control Office

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varduhi Petrosyan, MS, PHD, Principal Investigator — American University of Armenia Fund
Locations (1):
- School of Public Health, American University of Armenia Fund, Yerevan, Armenia

REFERENCES:
- [Background] Newell JN, Baral SC, Pande SB, Bam DS, Malla P. Family-member DOTS and community DOTS for tuberculosis control in Nepal: cluster-randomised controlled trial. Lancet. 2006 Mar 18;367(9514):903-9. doi: 10.1016/S0140-6736(06)68380-3. PMID 16546538
- [Background] Raza S, Sarfaraz M, Ahmad M. Practice of family and non-family based directly observed treatment for tuberculosis in Pakistan: A retrospective cohort study. The Health 2012; 3(2): 39-44
- [Background] Volmink J, Garner P. Directly observed therapy for treating tuberculosis. Cochrane Database Syst Rev. 2001;(4):CD003343. doi: 10.1002/14651858.CD003343. PMID 11687192
- [Background] Truzyan N, Harutyunyan T, Koshkakaryan M, Petrosyan V. Household TB Infection Control Pilot Project: Counseling for TB Patients and Their Family Members. American University of Armenia School of Public Health, Center for Health Services Research and Development, Yerevan, Armenia, 2013
- [Derived] Khachadourian V, Truzyan N, Harutyunyan A, Petrosyan V, Davtyan H, Davtyan K, van den Boom M, Thompson ME. People-centred care versus clinic-based DOT for continuation phase TB treatment in Armenia: a cluster randomized trial. BMC Pulm Med. 2020 Apr 25;20(1):105. doi: 10.1186/s12890-020-1141-y. PMID 32334553
- [Derived] Khachadourian V, Truzyan N, Harutyunyan A, Thompson ME, Harutyunyan T, Petrosyan V. People-centered tuberculosis care versus standard directly observed therapy: study protocol for a cluster randomized controlled trial. Trials. 2015 Jun 22;16:281. doi: 10.1186/s13063-015-0802-2. PMID 26093675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 12 March and 26 December 2014, we identified and contacted eligible TB patients from the intervention TB out-patient clinics as well as the control TB out-patient clinics.
Groups:
- Intervention Arm: The intervention included the following components: self-administered drug intake strategy, TB knowledge and socio-psychological counseling session, SMS text messages, phone calls, educational leaflet.
- Control Arm: Patients included in the control arm received traditional - clinical Directly Observed Therapy (DOT) as recommended by WHO.
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 194 | 198
Completed | 193 | 197
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 194 | 198 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (15.9) | 47.8 (14.9) | 46.8 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 48 | 87
  Male | 155 | 150 | 305

OUTCOME MEASURES:

1. Primary Outcome: TB Treatment Success Rates Defined by the World Health Organization (WHO)
Description: The sum of cured (TB patients with bacteriologically confirmed TB at the beginning of treatment who were smear- or culture-negative in the last month of treatment and on at least one previous occasion) and treatment completed (TB patients who completed treatment without evidence of failure but with no record to show that sputum smear or culture results in the last month of treatment and on at least one previous occasion were negative,either because tests were not done or because results are unavailable).
Time Frame: Patients were followed for the duration of ambulatory phase of treatment, an average of 4.2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 198 | 194
Participants | 184 | 176

2. Secondary Outcome: Knowledge About TB Infection
Description: Knowledge about TB infection will be measured by surveys
Time Frame: At baseline and upon completion of the treatment (an expected average of 4.5 months after starting the ambulatory phase of the treatment)
Reporting Status: Not Posted

3. Secondary Outcome: Stigma Level Towards TB Patients
Description: Stigma level towards TB patients will be measured by surveys
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: Family Support Towards TB Patients
Description: Change in family support towards TB patients will be measured by surveys
Time Frame: as for outcome 2
Reporting Status: Not Posted

5. Secondary Outcome: TB Treatment Adherence
Description: TB treatment adherence will be measured by surveys
Time Frame: as for outcome 2
Reporting Status: Not Posted

6. Secondary Outcome: Depression Status of TB Patients
Description: Depression status of TB patients will be measured by surveys
Time Frame: as for outcome 2
Reporting Status: Not Posted

7. Secondary Outcome: Quality of Life of TB Patients
Description: Quality of life of TB patients will be measured by surveys
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout the study period (average 4.2 months)
Arm/Group | Intervention Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 3/194 | 3/198
Other Adverse Events (participants affected / at risk) | 0/194 | 0/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=194) | Control Arm (N=198)
Death (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes